CLINICAL TRIAL: NCT07389265
Title: CAPRI-3 GOIM Study: Phase 3 Clinical Study to Evaluate the Use of Continuing Cetuximab Treatment Beyond First Line Progression in Molecular Selected Metastatic Colorectal Cancer Patients.
Brief Title: Continuation of Cetuximab Beyond First-Line Progression in Metastatic Colorectal Cancer
Acronym: CAPRI-3 GOIM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Fortunato Ciardiello, Principal Investigator, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPRI-3- GOIM Study
Record Dates: First submitted 2025-09-30; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Bevacizumab; Folfox protocol; Leucovorin; Fluorouracil; Oxaliplatin; Irinotecan

STUDY DESIGN:
Intervention Model Description: Patients will be randomized (1:1) into two arms:
  * Arm A: FOLFOX/FOLFIRI plus cetuximab
  * Arm B: FOLFOX/FOLFIRI plus bevacizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A Chemo-doublet (FOLFIRI or FOLFOX) + Cetuximab (Experimental): This arm is for participants with RAS/BRAF wild-type metastatic colorectal cancer who have progressed after first-line anti-EGFR therapy. They will receive a second-line chemotherapy regimen (either FOLFIRI or FOLFOX) in combination with cetuximab. The objective is to evaluate the efficacy of continuing cetuximab beyond progression.
  Interventions: Drug: Erbitux (Cetuximab); Drug: FOLFOX (Folinic acid + Fluorouracil + Oxaliplatin); Drug: FOLFIRI (5-Fluorouracil, Folinic acid, Irinotecan)
- ARM B Chemo-doublet (FOLFIRI or FOLFOX) + Bevacizumab (Active Comparator): This arm is for participants with RAS/BRAF wild-type metastatic colorectal cancer who have progressed after first-line anti-EGFR therapy. They will receive a second-line chemotherapy regimen (either FOLFIRI or FOLFOX) in combination with bevacizumab. This arm serves as the control group to compare the outcomes with the experimental arm.
  Interventions: Drug: Bevacizumab; Drug: FOLFOX (Folinic acid + Fluorouracil + Oxaliplatin); Drug: FOLFIRI (5-Fluorouracil, Folinic acid, Irinotecan)

INTERVENTIONS:
Drug: Erbitux (Cetuximab) — This is an anti-EGFR monoclonal antibody administered in combination with chemotherapy. The dose is 500 mg/m² administered every 14 days as a 120-minute intravenous infusion on cycle 1 day 1, infusion rate not faster than 5mg/min.
  Arms: ARM A Chemo-doublet (FOLFIRI or FOLFOX) + Cetuximab
Drug: Bevacizumab — This is an anti-VEGF monoclonal antibody used as an active comparator in the control arm of the study. The dose is 5 mg/kg of body weight, administered every 14 days
  Arms: ARM B Chemo-doublet (FOLFIRI or FOLFOX) + Bevacizumab
Drug: FOLFOX (Folinic acid + Fluorouracil + Oxaliplatin) — This is a standard chemotherapy regimen containing irinotecan, fluorouracil, and folinic acid. It is used as the backbone chemotherapy in both study arms.
  The dose includes 200 mg/m2 L-folinic acid given concurrently with 85 mg/ m² oxaliplatin over 2 h IV, followed by a 400 mg/ m² IV bolus of fluorouracil followed by 2400 mg/ m² fluorouracil IV infusion every 14 days.
Drug: FOLFIRI (5-Fluorouracil, Folinic acid, Irinotecan) — This is a standard chemotherapy regimen containing folinic acid, oxaliplatin, and fluorouracil. It is used as the backbone chemotherapy in both study arms.
  The dose includes 200 mg/m2 L-folinic acid given concurrently with 180 mg/ m² irinotecan over 1.30 h IV infusion, followed by a 400 mg/ m² IV bolus of fluorouracil followed by 2400 mg/ m² fluorouracil IV infusion over 46 h every 14 days.

SUMMARY:
The goal of this Phase 3 clinical trial is to evaluate whether continuing cetuximab treatment beyond first-line progression can improve outcomes in patients with metastatic colorectal cancer whose tumors are RAS and BRAF wild-type. The study will compare the effectiveness of chemotherapy given together with cetuximab versus chemotherapy given together with bevacizumab. Researchers aim to determine whether cetuximab continuation improves tumor response, progression-free survival, overall survival, and safety in this patient population.

Eligible participants are adults with metastatic colorectal cancer who have previously responded to first-line treatment with chemotherapy combined with an anti-EGFR antibody. Before starting therapy, patients will undergo molecular testing using liquid biopsy to confirm tumor characteristics. They will then receive chemotherapy with either cetuximab or bevacizumab every two weeks, and their disease will be monitored regularly with CT or MRI scans, laboratory tests, and clinical evaluations. During the study, patients will also provide biological samples for translational research.

This trial will enroll about 360 patients across sites in Italy and Spain and is designed to provide new evidence on whether cetuximab continuation beyond first-line treatment can offer a meaningful clinical benefit compared with standard therapy.

DETAILED DESCRIPTION:
Metastatic colorectal cancer (mCRC) is one of the most common and lethal cancers worldwide. Despite progress with chemotherapy and targeted therapies, many patients experience disease progression after first-line treatment. In recent years, drugs targeting the Epidermal Growth Factor Receptor (EGFR), such as cetuximab, have shown significant benefit in patients with RAS and BRAF wild-type tumors. However, it remains unclear whether continuing cetuximab beyond progression, while changing the chemotherapy backbone, can provide additional benefit compared to switching to an alternative targeted treatment.

The CAPRI-3 study is a randomized, multicenter, open-label Phase 3 clinical trial designed to address this question. The study will enroll approximately 360 adult patients with metastatic colorectal cancer in Italy and Spain. All participants must have tumors that are RAS and BRAF wild-type, as well as PIK3CA and EGFR extracellular domain wild-type and HER2 non-amplified, as determined by next-generation sequencing on liquid biopsy at the time of screening. Eligible patients will have previously received a first-line regimen with chemotherapy plus an anti-EGFR antibody (cetuximab or panitumumab) and achieved either a complete or partial response, or prolonged stable disease, before disease progression.

Patients will be randomized in a 1:1 ratio to receive a standard chemotherapy doublet (FOLFOX or FOLFIRI, depending on the regimen used in the first line) combined either with cetuximab (experimental arm) or with bevacizumab (control arm). Treatment will be continued until disease progression, unacceptable toxicity, or withdrawal of consent. Tumor response will be assessed according to RECIST 1.1 criteria by independent central review.

The primary endpoint of the study is objective response rate (ORR). Secondary endpoints include progression-free survival (PFS), overall survival (OS), and safety profile assessed according to NCI CTCAE version 5.0. Exploratory objectives include biomarker and translational research, involving the collection and analysis of tumor tissue, blood, and stool samples to better understand resistance mechanisms and the role of the gut microbiome in treatment response.

This study builds on promising results from the earlier CAPRI and CAPRI-2 trials, which suggested that continuing cetuximab in second-line therapy may improve patient outcomes. If successful, CAPRI-3 could establish cetuximab continuation beyond first-line progression as a new treatment option for a large proportion of molecularly selected patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of colorectal adenocarcinoma.
2. Diagnosis of metastatic disease.
3. Efficacy of a first line therapy containing anti-EGFR drug with a major response achieved (i.e. complete or partial response according to RECIST criteria v1.1) or a prolonged (at least 6 months) stable disease.
4. Progression to first line therapy.
5. RAS and BRAF wild-type status of FFPE analysis of primary colorectal cancer and/or related metastasis.
6. RAS (NRAS and KRAS exon 2,3 and 4), BRAFV600E, PIK3CA, EGFR ECD wild-type and HER2 not amplified in liquid biopsy at the time of screening (according to NGS, Foundation/Roche).
7. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST criteria, vers.1.1).
8. Male or female patients ≥ 18 years of age.
9. ECOG Performance Status 0-1.
10. Adequate bone marrow, liver and renal function assessed within 14 days before starting study treatment as defined by the following parameters:

    Bone marrow:
    * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
    * Hemoglobin (Hgb) ≥ 9 g/dL
    * Platelets ≥ 100 x 109/L

    Liver function:

    • Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and ALT (SGPT) ≤ 2.5 x ULN, except in patients with tumor involvement of the liver who must have AST and ALT ≤ 5 x ULN

    Renal function:

    • Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50 mL/min
11. If female and of childbearing potential*, have a negative result on a pregnancy test performed a maximum of 7 days before initiation of study treatment.

    *A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
12. If female and of childbearing potential, or if male, agreement to use adequate contraception (e.g., abstinence, intrauterine device, oral contraceptive, or double-barrier method), during the study and until at least 6 months after last dose of study treatment administration, based on the judgment of the Investigator or a designated associate.
13. Signed informed consent obtained before screening.

Exclusion Criteria:

1. Any contraindication to the use of cetuximab, bevacizumab, Irinotecan, 5-FU, oxaliplatin, folic acid.
2. Active uncontrolled infections, active disseminated intravascular coagulation or history of interstitial lung disease.
3. Past or current history of malignancies other than colorectal carcinoma, except for curatively treated basal and squamous cell carcinoma of the skin cancer or in situ carcinoma of the cervix.
4. Pregnancy (exclusion to be ascertained by a beta hCG test).
5. Breastfeeding.
6. Fertile women (<2 years after last menstruation) and men of childbearing potential not willing to use effective means of contraception.
7. Myocardial infarction, unstable angina pectoris, balloon angioplasty (PTCA) with or without stenting within the past 12 months before inclusion in the study, Grade III or IV heart failure (NYHA classification).
8. Cardiac arrhythmias requiring anti-arrhythmic therapy, with the exception of beta blockers or digoxin.
9. Medical or psychological impairments associated with restricted ability to give consent or not allowing conduct of the study.
10. Participation in a clinical study or experimental drug treatment within 30 days prior to study inclusion or during participation in the study.
11. Known or clinically suspected brain metastases.
12. History of acute or subacute intestinal occlusion or chronic inflammatory bowel disease or chronic diarrhea.
13. Severe, non-healing wounds, ulcers or bone fractures.
14. Marked proteinuria (nephrotic syndrome).
15. Known DPD deficiency (specific screening not required).
16. Known history of alcohol or drug abuse.
17. A significant concomitant disease which, in the investigating physician's opinion, rules out the patient's participation in the study.
18. Absent or restricted legal capacity.
19. Patients with known dMMR or MSI-H tumors who are eligible for approved immune checkpoint inhibitor therapy will be excluded from the trial, unless ICI therapy is contraindicated or declined by the patient. This ensures alignment with current standard of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, or study completion whichever came first, assessed until 48 months.
  The primary outcome is the Objective Response Rate, which will be evaluated according to the RECIST criteria 1.1. The study aims to determine if the continuous use of cetuximab in the experimental arm results in a superior Response Rate compared to the control arm with bevacizumab.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization (Day 0) until death from any cause, assessed through study completion (up to 36 months of survival follow-up)
  Time from randomization until death due to any cause. Patients alive at last follow-up will be censored at that date.
Progression-Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months from last patient randomized.
  Time from randomization until the date of first documented disease progression, as assessed by central independent review according to RECIST 1.1 criteria, or death from any cause, whichever occurs first.
Safety Profile: Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From first treatment administration until 30 days after the last dose.
  The safety profile of the trial drugs as measured by the incidence of AEs, SAEs, clinical laboratory assessments, vital signs, physical examination, ECG parameters, and ECOG PS.

CONTACTS AND LOCATIONS:
Overall Officials: Fortunato Ciardiello, Principal Investigator — A.O.U. dell'Università degli studi della Campania "Luigi Vanvitelli"
Locations (41):
- Italy (30):
  - A.O.U. Ospedali Riuniti, Ancona
  - AORN S. Giuseppe Moscati, Avellino
  - Centro di Riferimento Oncologico (C.R.O.) IRCCS, Aviano
  - IRCCS Istituto Tumori "Giovanni Paolo II", Bari
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Ospedale IRCCS 'Saverio de Bellis', Castellana Grotte
  - Nome EnteA.R.N.A.S. Garibaldi - P.O. Garibaldi-Nesima, Catania
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro
  - A.O.U. Careggi, Florence
  - P.O. 'Vito Fazzi', Lecce
  - Istituto Romagnolo per lo Studio dei Tumori 'Dino Amadori', Meldola
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Casa di Cura Villa Maria, Mirabella Eclano
  - A.O.U. dell'Università degli studi della Campania 'Luigi Vanvitelli', Napoli
  - A.O.U. Federico II, Napoli
  - IRCCS I.N.T. 'Fondazione G. Pascale', Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - ARNAS Civico - Di Cristina-Benfratelli - P. O. 'Civico e Benfratelli', Palermo
  - Casa di cura Macchiarella, Palermo
  - A.O.U. Pisana, Pisa
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia
  - Fondazione Policlinico Universitario 'Agostino Gemelli' IRCCS, Roma
  - IRCCS Istituto clinico Humanitas, Rozzano
  - Fondazione IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - A.O.U. Sassari, Sassari
  - Ospedale San Giuseppe Moscati, Statte
  - A.O. 'Pia Fondazione Cardinale G.Panico', Tricase
  - IRCCS Ospedale Sacro Cuore Don Calabria, Veneto
- Spain (11):
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona
  - Hospital General Universitario Santa Lucía, Cartagena
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Instituto Catalán de Oncología. Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario Marqués de Valdecilla, Santander